CLINICAL TRIAL: NCT04673396
Title: Phase I Clinical Study for Evaluation of Pharmacokinetic, Safety, Tolerance of Norcantharidin Lipid Microsphere for Injection in Patients With Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Nuokangda Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DXNCTD2019001
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumor
Keywords: Norcantharidin Lipid Microsphere For Injection; Pharmacokinetics; Safety; Tolerance
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Single center, open, non-randomized trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tolerance test (Experimental): The design is based on 3+3 dose escalation: three subjects were enrolled in each dose group, administered once a day for 2 weeks, and were observed for 7 days after withdrawal. If dose-limiting toxicity (DLT) was not observed, the dose was incresed to the next dose group. If dose-limiting toxicity (DLT) was found in 2 or more patients in a given dose group, the climbing test was terminated and the dose was reduced by 1 dose. If there were only three subjects, three more subjects were observed, so that the MTD dose group had at least six evaluable subjects.If DLT occurs in 1 patient in a given dose group, 3 more subjects should be added to that dose group. If DLT occurs in 1 or more of these 3 subjects, the climb will be stopped and the dose group will be reduced by 1 dose group. If there are only 3 subjects, 3 more subjects will be observed, so that at least 6 patients in the MTD dose group can be evaluated.
  Interventions: Drug: Norcantharidin Lipid Microsphere for Injection
- Pharmacokinetic studies (Experimental): At the same time of tolerance test, blood PK sampling was performed. At the end of the tolerance test in each group, on the premise of good safety, and after evaluation by the researchers, additional cases were selected from the three dose groups (low, medium and high) for pharmacokinetic study, so as to ensure that at least 8 patients could be evaluated for PK in each group.
  Interventions: Drug: Norcantharidin Lipid Microsphere for Injection
- Comparative Study (Active Comparator): It is planned to select the 20mg dose of norcantharidin sodium for injection to carry out pharmacokinetic study of 8 cases. The specific research design will be formulated after the tolerance and pharmacokinetic test of norcantharidin lipid microsphere injection is completed.
  Interventions: Drug: Norcantharidin Lipid Microsphere for Injection; Drug: Sodium Demethylcantharidate Injection

INTERVENTIONS:
Drug: Norcantharidin Lipid Microsphere for Injection — The test drug was added to 5% glucose injection to a final volume of 250 mL，and administered by instillation at a rate of 200 mL/h.
  This product can be used alone or in combination with chemotherapy, and the dosage and time of administration vary with the chemotherapy regimen.
  Other Names: Tolerance,and Pharmacokinetic study
Drug: Sodium Demethylcantharidate Injection — Dissolve the reference drug with appropriate amount of sterile water for injection, and add 250 mL of 5% glucose injection for slow dripping.
  Other Names: Comparative Pharmacokinetic Studies
  Arms: Comparative Study

SUMMARY:
This study was designed as a single-center, open, non-randomized trial.

DETAILED DESCRIPTION:
In this study, patients with locally advanced or metastatic solid tumors were enrolled for a tolerance test and a pharmacokinetic study. The dosage increment principle of 3+3 was adopted. At the end of the tolerance test, 3 dose groups (low, medium and high) were selected to conduct pharmacokinetic studies after evaluation by the researchers on the premise of good safety, and at least 8 patients were included in each group for PK study (at least 8 patients in each group could be evaluated for PK ).

After the end of the experimental drug tolerance and pharmacokinetics study, the safety and pharmacokinetics of single dose administration were compared with that of sodium norcantharidate for injection in the dose range of clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, regardless of gender.
2. Condition body mass index (BMI) = Weight (kg)/Height 2 (m2), the body mass index is in the range of 18-28 (Including the cut-off value).
3. Patients with locally advanced or metastatic solid tumors that have been clearly diagnosed by histology/cytology, patients whose condition is stable after standard treatment, or those who have failed standard treatment.
4. According to the Eastern Cooperative Oncology Group (ECOG) score of 0 to 2, the estimated survival time is ≥ 3 months.
5. It has sufficient organ and bone marrow functions, defined as follows:

   1. Blood routine: white blood cell count (WBC) ≥ 4.0 × 109/L; neutrophil count (NEUT) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 100 × 109/L; hemoglobin concentration ≥ 9.0 g/ dL;
   2. Liver function: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); for patients with liver cancer or liver metastases, ALT and AST ≤ 5 times ULN; Total bilirubin (TBIL) ≤ 1.5 × ULN;
   3. Renal function: blood creatinine (CREA) ≤ 1.5 × ULN;
   4. Heart function: LVEF ≥ 50%.
6. Those who have used chemotherapeutics in the past need to stop the drug for more than 4 weeks (mitomycin or nitrosourea, need to stop for more than 6 weeks); have received surgery, molecular targeted therapy, and anti-tumor indications with Chinese medicine Those who need treatment should end at least 4 weeks, and those who have received palliative radiotherapy need more than 4 weeks of treatment.
7. Any toxicity associated with previous anti-tumor treatments must have been restored to ≤ Grade 1 (except for hair loss).
8. During the study period and within 3 months after the end of the administration, subjects with fertility (whether male or female) must receive effective contraceptive measures.
9. With my consent and signed an informed consent form by myself or my legal representative.

Exclusion Criteria:

1. Suffer from any clinically significant cardiovascular and cerebrovascular diseases within 3 months before taking the trial drug, including but not limited to myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, congestive heart failure, Cerebrovascular accident (including transient ischemic attack).
2. There is NCI-CTCAE grade ≥ grade 2 arrhythmia, any grade of atrial fibrillation that is not controlled, or the ECG found at the time of screening that the QT interval (QTc) for two consecutive corrections> 480ms.
3. Any drug that may prolong the QTc interval or induce torsade de pointes ventricular tachycardia is required within 14 days before the first use of the test drug or during treatment.
4. History of allergic diseases and severe drug allergy.
5. Patients with uncontrolled tumor brain metastases with clinical symptoms.
6. Patients with severe infections (including but not limited to progressive or active infections) (for example, intravenous infusion of antibiotics, antifungal or antiviral drugs, etc.).
7. Patients with severe medical diseases, such as cardiac dysfunction of grade II and above (NYHA standard), ischemic heart disease (such as myocardial infarction or angina), congestive heart failure and other cardiovascular diseases, poorly controlled diabetes (Fasting blood glucose ≥10mmol/L), poorly controlled hypertension (systolic blood pressure>150mmHg and/or diastolic blood pressure>100mmHg).
8. Those who have bleeding tendency or are receiving thrombolysis or anticoagulation therapy.
9. Active hepatitis (hepatitis B, hepatitis C) or known HIV infection.
10. Other systemic anti-tumor treatments may be accepted during the study period.
11. A clear history of neurological or mental disorders, including epilepsy or dementia.
12. Have bad habits such as drug and alcohol abuse. Alcoholism refers to drinking behaviors of 4 or more times within about 2 hours. One-time drinking refers to drinking 150ml of wine, 350ml of beer, or 50ml of 80% liquor (or equivalent to the alcohol content).
13. Women during pregnancy or lactation.
14. Those who have received other drug clinical research within 1 month before the study.
15. Other situations where the researcher thinks it is inappropriate to participate in this research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | ±1 minute
  Obtain directly according to the measured data of blood drug concentration-time.
AUC 0-t | ±1 minute
  The area under the curve from the time of administration to the lowest detectable blood concentration: calculated by the linear trapezoidal rule.
AUC 0-∞ | ±1 minute
  Area under the curve from administration to extrapolation to infinity: AUC0-∞=AUC0-t+Ct/λz, Ct is the last measurable concentration, and λz is the elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, Ph.D, Principal Investigator — The First Affiliated Hospital, China Medical University
Locations (1):
- The First Affiliated Hospital, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No